CLINICAL TRIAL: NCT03204006
Title: Attenuation of Hemodynamic Response to Laryngoscopy and Endotracheal Intubation With Single Dose of Dexmedetomidine in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman A. Ismail, Lecturer of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 01003060483
Record Dates: First submitted 2017-06-26; First posted 2017-06-29 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Stress Response During Laryngoscopy Intubation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Active Comparator): 35 patients will receive dexmedetomidine 0.5 µg/kg was administered intravenously using a syringe pump over 10 min sterile saline pre-induction of anesthesia.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): 35 patients will receive sterile saline 0.5 µg/kg was administered intravenously using a syringe pump over 10 min pre-induction of anesthesia.
  Interventions: Drug: sterile saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine preinduction
  Arms: Dexmedetomidine group
Drug: sterile saline — normal saline preinduction
  Arms: Control group

SUMMARY:
Attenuation of Hemodynamic Response to Laryngoscopy and Endotracheal Intubation With Single Dose of Dexmedetomidine in Hypertensive Patients.

ELIGIBILITY:
Inclusion Criteria:

* - Age group 20-60 years
* ASA grade 1 and 2
* control hypertensive patients.

Exclusion Criteria:

* - Consent not given
* ASA Grade 3 and 4
* history of myocardial ischemia or infarction, or had an abnormal ECG on admission to the hospital
* Patients with cardiovascular, pulmonary, hepatic, and renal disease.
* Patients on B blockers.
* patients with difficult airway; laryngoscopy and intubation time more than 20 s, or requiring more than two attempts will be exclude from the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2020-03-08 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
heart rate | through first 15 min post-induction of anesthesia

SECONDARY OUTCOMES:
systolic blood pressure | through first 15 min post-induction of anesthesia
diastolic blood pressure | through first 15 min post-induction of anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt